CLINICAL TRIAL: NCT05585775
Title: Affective Executive Functioning as a Mechanism of Treatments for Depression Symptoms
Brief Title: Mood and Thought Process Study
Acronym: MAT Process
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Morganne Kraines, Research Psychologist, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2110-001; K23AT011388-01A1 (NIH)
Record Dates: First submitted 2022-10-11; First posted 2022-10-19 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Depression in Remission; Depressive Symptoms; Depression
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): MBCT classes are comprised of weekly, 2.5-hour classes in which participants learn cognitive therapy techniques and practice meditation exercises. Participants will complete group and/or individual orientation to MBCT with the MBCT instructor, 1-2 weeks prior to the first scheduled MBCT class. Additionally, MBCT requires 45-minutes of daily home practice, and a full day, 8-hour silent meditation retreat. MBCT classes are delivered via the protocol and curriculum developed by the MBCT founders. Participants randomized to MBCT will receive 8-weeks of MBCT classes.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Wellness for Wellbeing (Active Comparator): Wellness for Wellbeing will serve as the active control for MBCT. Participants randomized to Wellness for Wellbeing will receive 1-hour group delivered classes, once per week, for 8-weeks. Participants will receive an orientation to Wellness for Wellbeing 1-2 weeks prior to the first class. Classes will be delivered by a research therapist. Topics for Wellness for Wellbeing include: nutrition, caffeine, preventing cancer, diabetes, heart health, sleep, being a smart patient, and complementary and alternative medicine. Wellness for Wellbeing classes are interactive and do not include components designed to impact affective cognition in any way. Because participants may have varying levels of health literacy, the research therapist tailors presentation of the material to the participants' level of knowledge of the topic. Information presented in Wellness for Wellbeing is regularly updated with current health guidelines.
  Interventions: Behavioral: Wellness for Wellbeing

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — MBCT classes are comprised of weekly, 2.5-hour classes in which participants learn cognitive therapy techniques and practice meditation exercises. Participants will complete group and/or individual orientation to MBCT with the MBCT instructor, 1-2 weeks prior to the first scheduled MBCT class. Additionally, MBCT requires 45-minutes of daily home practice, and a full day, 8-hour silent meditation retreat. MBCT classes are delivered via the protocol and curriculum developed by the MBCT founders. Participants randomized to MBCT will receive 8-weeks of MBCT classes.
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Behavioral: Wellness for Wellbeing — Wellness for Wellbeing will serve as the active control for MBCT. Participants randomized to Wellness for Wellbeing will receive 1-hour group delivered classes, once per week, for 8-weeks. Participants will receive an orientation to Wellness for Wellbeing 1-2 weeks prior to the first class. Classes will be delivered by a research therapist. Topics for Wellness for Wellbeing include: nutrition, caffeine, preventing cancer, diabetes, heart health, sleep, being a smart patient, and complementary and alternative medicine. Wellness for Wellbeing classes are interactive and do not include components designed to impact affective cognition in any way. Because participants may have varying levels of health literacy, the research therapist tailors presentation of the material to the participants' level of knowledge of the topic. Information presented in Wellness for Wellbeing is regularly updated with current health guidelines.
  Arms: Wellness for Wellbeing

SUMMARY:
The primary objective for this project is to test whether affective executive functioning is a mechanism of action of mindfulness-based cognitive therapy and Wellness for Wellbeing. The main questions it aims to answer are:

1. Test the effect of MBCT vs. Wellness for Wellbeing on affective inhibition (i.e., emotionally valenced inhibition as measured via the affective Go/No Go task) using an RCT.
2. Test the effect of MBCT vs. Wellness for Wellbeing on (a) affective updating and (b) affective shifting. Outcomes will be measured with the affective n-Back and the affective Internal Switching Task, respectively.

3a) The investigators will examine whether depression symptom severity co-varies with change in affective executive functioning (i.e., affecting inhibition, shifting, and updating) over time. 3b) The investigators will examine whether compliance with treatment protocol (e.g., number of classes attended, amount of home practice) predicts endpoint executive functioning.

Participants will complete surveys, interviews, and computer tasks, and will be randomized to either Mindfulness-Based Cognitive Therapy or Wellness for Wellbeing.

DETAILED DESCRIPTION:
Mindfulness-Based Cognitive Therapy (MBCT) is an efficacious treatment for patients with symptoms of depression. However, the processes by which MBCT achieves its outcomes are not well understood. Drawing on literature on basic cognitive functioning and cognitive biases in depression, this K23 will use a randomized controlled trial to test the effect of MBCT vs. Wellness for Wellbeing on affective inhibition (an important component of executive functioning (EF)), and a possible mechanism of action by which MBCT has an impact on depression symptoms. As a secondary aim, this project will also test the effect of MBCT vs. Wellness for Wellbeing on affective updating and affective shifting (two remaining components of EF). In exploratory analyses, the investigators will examine whether depression symptom severity covaries with change in affective EF (i.e., affective inhibition, shifting, and updating) overtime, and whether adherence to the treatment protocol predicts endpoint EF. To accomplish these goals, 76 adult participants with elevated depression symptoms will be recruited from the community and will be randomized to either an 8-week MBCT course at the Mindfulness Center at Brown University or an 8-week Wellness for Wellbeing Class. Participants will complete validated computer-based tasks of affective EF at 4-assessments, 1 before, 2 during, and 1 after, the 8-week MBCT or Wellness for Wellbeing programs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years or older
2. English fluency in order to complete study procedures
3. Normal vision or corrected to normal vision
4. QIDS score ≥ 5 and ≤ 15 to include individuals with elevated, but not severe symptoms of depression
5. No presence of psychotic symptoms that interfere with functioning
6. No current hazardous alcohol or drug use
7. No previous experience with mindfulness-based treatment (i.e., enrollment in MBSR or MBCT previously)
8. No current symptoms of mania indicative of a manic episode
9. No current cognitive impairment
10. No history of a formally diagnosed learning disability in reading, intellectual disability or other developmental disorder
11. No history of a neurologic illness affecting cognition
12. If on psychiatric medications, no change in medications for at least 4 weeks
13. If in psychotherapy, no change in therapy status for at least 4 weeks

Exclusion Criteria:

Exclusion criteria include: (a) presence of psychotic symptoms that interfere with one's ability to function as determined by the SCID-5 Psychotic Screening Module; (b) current hazardous alcohol or drug use as indicated by a score of >10 for men and women on the AUDIT and the DUDIT for cannabis use, and >6 for men and women on the DUDIT for all other drugs (everything but cannabis), (c) change in psychiatric drug prescription within 4 weeks; (d) started psychotherapy or other psychiatric treatment within the past 4 weeks; (e) current suicide ideation or behavior which requires urgent intervention due to safety concerns; (f) Previous enrollment in MBCT or MBSR; (g) symptoms of mild cognitive impairment as indicated by a score of <26 on the MoCA; (h) formally diagnosed learning disability, intellectual disability, or other developmental disorder; (i) history of neurologic illness affecting cognition; (j) current symptoms indicative of a manic episode per the SCID-5 Mood Disorders Module.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Affective Go/No-Go | 10-week
  This task requires utilizing inhibition to respond to word features (i.e., normal vs. italicized font) rather than word content. In this task, participants are told to respond (via key press) when a go stimulus (i.e., normal text) is presented and to withhold their response when a no-go stimulus (i.e., italicized text) is presented. words are negatively valenced (e.g., hate, sad) or positively valenced (e.g., terrific, win). Conditions are matched on word length and frequency of use in the English language.
Emotional n-back | 10-week
  Updating will be measured via the n-Back Task. Individuals are presented words on a computer screen, and are asked to indicate (via key press), whether the current word is the same or different from the word presented n times back. The investigators will be using 2-back trials, as these trials are not too difficult so that participants become frustrated, yet engage updating processes. The affective version of the task will be an adapted affective n-back task in which individuals are presented with negative and positive words, and asked to indicate via key press whether the word n-trials back matches the valence (positive or negative) of the current word.
Affective Internal Switching Task | 10-week
  Shifting will be measured via the Internal Switching Task (IST). Participants are presented with one word on the computer screen at a time, and are asked to keep a silent mental count of how many words they see from two semantic categories (i.e., positive affective words and negative affective words). Participants are instructed to press the spacebar when they have updated their mental count and are ready for the next word. Participants are asked to keep a mental count of how many positive and how many negative words appear in each category, and press the spacebar when they have updated their mental count.
Depression Symptoms | 10-week
  Participants will complete the 16-item Quick Inventory of Depression Symptoms (Self-Report) measure assessing depression symptoms and associated symptoms.

SECONDARY OUTCOMES:
Attention Control Scale | 10-week
  Self-report measure of attention control
Positive and Negative Affect Scale | 10-week
  Self-report measure of affect
Five Factor Mindfulness Scale | 10-week
  Self-report measure of mindfulness
Patient Health Questionnaire-9 | 10-week
  Self-report measure of depression symptoms
Ruminative Response Scale | 10-week
  Self-report measure of rumination
Generalized Anxiety Disorder -7 | 10-week
  Self-report measure of anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Morganne Kraines, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Because data from this project will be completely de-identified and our sample will not be easily identifiable, data will be made available upon request to other researchers without cost to researchers or analysts.